CLINICAL TRIAL: NCT06309459
Title: Carbonic Anhydrase IX Enzyme in Triple Negative Breast Carcinoma: Relationship With Prognostic Factors and Response to Neoadjuvant Chemotherapy
Brief Title: Carbonic Anhydrase IX Enzyme in Triple Negative Breast Carcinoma
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: IRB 2023/04-34
Record Dates: First submitted 2024-01-10; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Triple Negative Breast Cancer; Carbonic Anhydrase IX
Keywords: Triple negative breast carcinoma; Carbonic anhydrase IX; Treatment effect; Ki67 proliferation index
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Postop mastectomy pathologic materials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Staining: CA IX is a transmembrane protein, it exhibits cytoplasmic membrane staining. Immunohistochemically positive cells were graded as Low staining if they constituted <10% of the total.
  Interventions: Diagnostic Test: Carbonic anhydrase staining levels
- High Staining: CA IX is a transmembrane protein, it exhibits cytoplasmic membrane staining. Immunohistochemically positive cells were graded as high staining if they constituted ≥ 10%
  Interventions: Diagnostic Test: Carbonic anhydrase staining levels

INTERVENTIONS:
Diagnostic Test: Carbonic anhydrase staining levels — CA IX is a transmembrane protein, it exhibits cytoplasmic membrane staining. Immunohistochemically positive cells were graded as Low staining if they constituted <10% of the total and high staining if they constituted ≥ 10% (15).

SUMMARY:
Triple-negative breast carcinoma is characterized by the absence of estrogen receptors, progesterone receptors, and HER2/neu receptors. Carbonic anhydrase IX (CA IX) is a tumor-associated cell surface glycoprotein that is involved in adaptation to hypoxia-induced acidosis and plays a role in cancer progression. This study aimed to investigate CA IX expression in TNBC and its relationship with treatment effect.

DETAILED DESCRIPTION:
Tru-cut biopsy materials, sent to our hospital pathology laboratory between August 2018 and May 2023, will be examined. Invasive carcinoma cases will be evaluated according to estrogen, progesterone, and HER 2 receptor levels. Triple-negative tumor cases were isolated and those cases who underwent breast resection in our hospital after receiving neoadjuvant chemotherapy (Adriamycin, cyclophosphamide, and then paclitaxel for 4 cycles) were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Triple-negative mastectomy cases
* Patients whose data can be available
* Patients who were operated in our hospital

Exclusion Criteria:

* Younger than 18 years
* Not triple negative mastectomy cases
* Patients with missing data
* Patients who were operated in another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Triple Negative Breast Cancer cases who were operated in Elazığ Fethi Sekin SUAM
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Poor prognostic factors in patients with TNBC | 2018-2023
  Higher staining CA IX levels (≥ 10%) in TNBC patients' pathological specimens is a poor prognostic factor
The treatment success with inhibiting the CA IX enzyme levels' effectiveness | 2018-2023
  Treatment success in TNBC patients by evaluating changes in CA IX staining levels

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakherad H, Ghasemi F, Hosseindokht M, Zare H. Nanobodies; new molecular instruments with special specifications for targeting, diagnosis and treatment of triple-negative breast cancer. Cancer Cell Int. 2022 Aug 6;22(1):245. doi: 10.1186/s12935-022-02665-0. PMID 35933373
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Yin L, Duan JJ, Bian XW, Yu SC. Triple-negative breast cancer molecular subtyping and treatment progress. Breast Cancer Res. 2020 Jun 9;22(1):61. doi: 10.1186/s13058-020-01296-5. PMID 32517735
- [Background] Warburg O, Wind F, Negelein E. THE METABOLISM OF TUMORS IN THE BODY. J Gen Physiol. 1927 Mar 7;8(6):519-30. doi: 10.1085/jgp.8.6.519. No abstract available. PMID 19872213
- [Background] Carroll CP, Bolland H, Vancauwenberghe E, Collier P, Ritchie AA, Clarke PA, Grabowska AM, Harris AL, McIntyre A. Targeting hypoxia regulated sodium driven bicarbonate transporters reduces triple negative breast cancer metastasis. Neoplasia. 2022 Mar;25:41-52. doi: 10.1016/j.neo.2022.01.003. Epub 2022 Feb 9. PMID 35150959
- [Background] Lee P, Chandel NS, Simon MC. Cellular adaptation to hypoxia through hypoxia inducible factors and beyond. Nat Rev Mol Cell Biol. 2020 May;21(5):268-283. doi: 10.1038/s41580-020-0227-y. Epub 2020 Mar 6. PMID 32144406
- [Background] Godet I, Doctorman S, Wu F, Gilkes DM. Detection of Hypoxia in Cancer Models: Significance, Challenges, and Advances. Cells. 2022 Feb 16;11(4):686. doi: 10.3390/cells11040686. PMID 35203334
- [Background] Gillies RJ, Brown JS, Anderson ARA, Gatenby RA. Eco-evolutionary causes and consequences of temporal changes in intratumoural blood flow. Nat Rev Cancer. 2018 Sep;18(9):576-585. doi: 10.1038/s41568-018-0030-7. PMID 29891961
- [Background] Wu Q, You L, Nepovimova E, Heger Z, Wu W, Kuca K, Adam V. Hypoxia-inducible factors: master regulators of hypoxic tumor immune escape. J Hematol Oncol. 2022 Jun 3;15(1):77. doi: 10.1186/s13045-022-01292-6. PMID 35659268